CLINICAL TRIAL: NCT01003756
Title: Preoperative Exercise in Patients Undergoing Total Hip or Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Allan Villadsen, MD, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: s-20090099
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Osteoarthritis
Keywords: Preoperative; Exercise; Joint Replacement; Hip; Knee
MeSH Terms: conditions — Osteoarthritis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- Knee Intervention (Experimental): Patients undergoing Total Knee Replacement. Exercise 8-10 weeks preoperatively
  Interventions: Other: Preoperative neuromuscular exercise
- Knee Control (No Intervention): Patients undergoing Total Knee Replacement. Receives standard instructions
- Hip Intervention (Experimental): Patient undergoing Total Hip Replacement. Exercise 8-10 weeks preoperatively
  Interventions: Other: Preoperative neuromuscular exercise
- Hip Control (No Intervention): Patients undergoing Total Hip Replacement. Receives standard instructions

INTERVENTIONS:
Other: Preoperative neuromuscular exercise — A neuromuscular exercise programme delivered 8-10 weeks preoperatively. The programme is developed in Lund, Sweden. A journal of this study is under peer-review
  Arms: Hip Intervention; Knee Intervention

SUMMARY:
This study is conducted in the Community Hospital in Svendborg (OUH Svendborg Sygehus) in collaboration with University of Southern Denmark and Odense University Hospital.

The overall purpose of this study is to evaluate the effects of preoperatively delivered neuromuscular exercise on self perceived physical function, pain and Quality of Life in patients undergoing total hip or knee replacement. Secondary area of interest is physical performance, muscle function, and level of physical activity.

The project will be conducted in two phases:

* A pilot project focusing on the logistics of the upcoming randomized controlled trial (RCT) and determination of test-retest reliability of specific muscle strength variables for the patients of interest
* A randomized and controlled trial where the intervention is preoperative neuromuscular exercise and the controls receive standard instructions.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective primary, unilateral total hip or knee replacement in Svendborg Community Hospital, Odense University Hospital, Denmark.
* Patients with osteoarthritis
* Age over 18

Exclusion Criteria:

* Not being able to read and understand Danish.
* Patients with co-morbidity diseases where a moderate level of physical exercise is contraindicated, e.g. severe heart disease and neurological deficits.
* Patients unable to attend intervention.
* Rheumatoid arthritis (RA). A history of or ongoing use of medication for RA or other inflammatory arthritis such as gold, methotrexate, plaquenil etc.
* Lack of wish to participate or unwillingness to sign an informed consent.
* Specific for hip patients: a history of severe sequelae due to congenital hip-dysplasia requiring specialized postoperative training. A history of femoral neck and trochanteric fracture.
* Patients planned to have bilateral joint replacement within same procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2009-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in self reported physical function. Assessed with KOOS/HOOS questionnaire subscale ADL Function | 3 month postoperative (primary endpoint)
  Further assessments: baseline, preoperative, 6 weeks postoperative and 1-year follow up

SECONDARY OUTCOMES:
Self reported pain. Assessed with KOOS and HOOS subscale on pain. | baseline, one week preop., 3 month postop.(primary endpoint) and a 1 year follow up
Self reported quality of life (Qol). Assessed with KOOS and HOOS sub scale quality of life | baseline, one week preop., 3 month postop.(primary endpoint) and a 1 year follow up
Self reported quality of life. Assessed with EQ5D questionnaire | baseline, one week preop., 3 month postop.(primary endpoint) and a 1 year follow up
Observed physical function. Assessed with performance measures: 20 meter walk, 5 chair stands timed and one leg knee bendings/30 sec | baseline, one week preop. and 3 month postop.
Muscle strength estimated as average muscle power for muscles of the hip and knee | baseline, 1 week preop. and 3 month postop

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Roos, Professor, PT, PhD, Study Chair — University of Southern Denmark; Allan Villadsen, MD, Principal Investigator — University of Southern Denmark
Locations (1):
- Dept. of Orthopedics Svendborg Community Hospital, Svendborg, Denmark

REFERENCES:
- [Derived] Fernandes L, Roos EM, Overgaard S, Villadsen A, Sogaard R. Supervised neuromuscular exercise prior to hip and knee replacement: 12-month clinical effect and cost-utility analysis alongside a randomised controlled trial. BMC Musculoskelet Disord. 2017 Jan 6;18(1):5. doi: 10.1186/s12891-016-1369-0. PMID 28061841
- [Derived] Villadsen A, Overgaard S, Holsgaard-Larsen A, Christensen R, Roos EM. Immediate efficacy of neuromuscular exercise in patients with severe osteoarthritis of the hip or knee: a secondary analysis from a randomized controlled trial. J Rheumatol. 2014 Jul;41(7):1385-94. doi: 10.3899/jrheum.130642. Epub 2014 Jun 15. PMID 24931956
- [Derived] Villadsen A, Overgaard S, Holsgaard-Larsen A, Christensen R, Roos EM. Postoperative effects of neuromuscular exercise prior to hip or knee arthroplasty: a randomised controlled trial. Ann Rheum Dis. 2014 Jun;73(6):1130-7. doi: 10.1136/annrheumdis-2012-203135. Epub 2013 May 9. PMID 23661494